CLINICAL TRIAL: NCT01854749
Title: S1 Combined With Cisplatin in Treatment of Recurrence/Metastasis of ESCC Open-label Single Center Phase II Clinical Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Chang Jian Hua, Deputy director of medical oncology, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S1- ESCC -CJH
Record Dates: First submitted 2013-05-10; First posted 2013-05-16 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: ESCC
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- S1 combined with cisplatin (Experimental)
  Interventions: Drug: S1 combined with cisplatin

INTERVENTIONS:
Drug: S1 combined with cisplatin

SUMMARY:
Assess the efficacy and safety of S1 combined with cisplatin in treatment of recurrence/metastasis of ESCC

ELIGIBILITY:
Inclusion Criteria

* Joined the study voluntarily and signed informed consent form;
* Age 18-75

  .Presence of at least one index lesion measurable by CT scan or MRI
* recurrence/metastasis of Esophageal carcinoma or gastroesophageal cancer confirmed by pathology
* No radiotherapy, chemotherapy or other treatments prior to enrollment
* PS ECOG 0-1
* Life expectancy of more than 3 months
* ANC≥2×109/L，PLT≥100×109/L，Hb≥90g/L

  * Cr≤1.0×UNL
  * TBIL≤1.25×UNL； ALT/AST≤2.5×UNL，with hepatic metastases ALT/AST≤5.0×UNL；AKP≤2.5×UNL

Exclusion Criteria:

* there is radical cure of the cancer

  * uncontrolled chronic diarrhea and esophageal obstruction
  * Neurological or mental abnormalities Influence of cognitive ability include central nervous system metastases
  * Severe complication(s), e.g.,uncontrolled active infection,myocardial infarction,hypertension,arrhythmia,stenocardia
  * Patient who has metastasis except cured skin basal cell carcinoma and carcinoma in situ of cervix
* accept other antitumor therapy •Female patients during their pregnant and lactation period, or patients without contraception

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2011-11; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | from the first cycle of treatment (day one) to two month after the last cycle

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer hospital Fudan University, Shanghai, Shanghai Municipality, China